CLINICAL TRIAL: NCT04910282
Title: Impact of COVID-19 on Quality of Life of Seniors With Eye Disease and Implementations to Improve Wellness
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 115875
Record Dates: First submitted 2021-05-31; First posted 2021-06-02 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Covid19; Eye Diseases
Keywords: Eye disease patients; Psychological stressors; COVID-19; Seniors
MeSH Terms: conditions — COVID-19; Eye Diseases; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eye Disease Patients: Patients with eye diseases age 65 and above will be included. Patients from the Ivey Eye Institute, St. Joseph's Health Care London, ON will be recruited in-person, based on inclusion and exclusion criteria.

SUMMARY:
The ophthalmology clientele is vulnerable in the context of the coronavirus disease 2019 (COVID-19) pandemic because of their age and comorbidities. Specifically, elderly patients aged 65 and above with glaucoma, age-related macular degeneration, or diabetic retinopathy require regular follow-ups and commonly suffer from additional comorbidities. Further, because of the proximity between the patient and health care personnel during ophthalmological examinations, the risk of infection during visits is significant. The delicate balance between the risk of exposure to COVID-19 and visual loss in delaying cases is a psychological stressor to both patients and clinicians.

A cross-sectional study accumulating the data of 425 patients aged 65 and above with various eye diseases will be conducted. Participants will be presented with a set of online questionnaires designed to collect data on health-related quality of life (HRQOL), vision-related quality of life (VRQOL), depression symptoms, anxiety, sleep quality, community integration, and their experience with tele-consultations. This study can help quantify the collateral impact of the COVID-19 beyond the direct impact of the virus, to improve future quality of care guidelines on non-COVID-19 conditions, and to help plan patient prioritization once restrictions are eased.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

COVID-19 is caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Like many healthcare departments, the department ophthalmology presents risk of COVID-19 infection. As a result, the present pandemic has led officials to rethink the management of patient lists and to restrict the patients to be assessed or to be operated based on the urgency of their condition in accordance with ministerial guidelines. A delay in visits might increase the risk of visual loss not only through the delay of necessary care, but also through an increase in non-adherence to treatment. Indeed, patients themselves might decide to interrupt their treatment or postpone their visit for fear of contracting the disease. There is concern not only about compliance to treatment, but also about accessibility issues to medications in high-demand and modifications of treatment protocols.

Elderly people aged 65 and above are commonly afflicted by many eye diseases with vision loss. Furthermore, during times of the COVID-19 pandemic, this population can be vulnerable to possible vision loss due to a delay of care.

As a result, it is being proposed to perform a cross-sectional study using a sample of patients from this population to gather information on follow-up and treatment delays associated with the pandemic's offloading measures as well as any adverse effects on visual acuity that have occurred during the pandemic. The evidence collected from this study could be translated into clinical practices helping to provide recommendations to adjust the response to the COVID-19 pandemic in ophthalmological management.

Visual loss, potentially due to the reasons that were mentioned above, can bring about depressive symptoms and deteriorate the quality of life (QOL). In the proposed study, the investigators have included questionnaires to assess the various stressors brought on during the COVID-19 pandemic such as fear of vision loss, health-related QOL, vision-related QOL, depression and anxiety symptoms, sleep quality, number of ER visits for deterioration of mental health. This evidence base collected from this study could, once again, be translated into clinical practices helping to provide recommendations to adjust the response to the COVID-19 pandemic in ophthalmological management.

STUDY AIM

Through a cross-sectional survey, the investigators aim to build an evidence base to provide decision-makers with high quality, timely, and relevant evidence and to translate this knowledge into clinical practices by providing real-time knowledge and recommendations to adjust the response to the COVID-19 pandemic in ophthalmological management.

STUDY OBJECTIVES AND HYPOTHESES

Primary objectives: To build an evidence base to provide decision-makers with high quality, timely, and relevant evidence and to translate this knowledge into clinical practices by providing real-time knowledge and recommendations to adjust the response to the COVID-19 pandemic in ophthalmological management.

Secondary objectives: Using a cross-sectional survey, the investigators will: 1) document the follow-up and treatment delays associated with the pandemic's offloading measures 2) determine whether any adverse effects on visual acuity occurred during the pandemic 3) determine the impact on mental health (e.g. fear of vision loss, health-related QOL, vision-related QOL, depression and anxiety symptoms, sleep quality, number of ER visits for deterioration of mental health) 4) determine the role and impact of virtual care (telemedicine, teleconsultation) in the state of the current pandemic and provide additional data for the long-term implementation of telemedicine in vision care.

METHODOLOGY

Study Design

A cross-sectional survey will be performed to gather the data required to build an evidence base to provide decision-makers with high-quality, timely, and relevant evidence, as well as to translate this knowledge into clinical practices.

Study Population and Setting

Patients from the Ivey Eye Institute, St. Joseph's Health Care London, ON will be recruited in-person, similar to the previous and ongoing research studies by the investigators, based on inclusion and exclusion criteria.

Recruitment

It is being hoped to complete recruitment within a year of receiving ethics approval. Based on previous experience, it is planned to recruit at an average rate of 4 participants/week in a staggered manner over a 9 to 10-month period.

Data Fidelity, and Management

Day-to-day Management of the Study

The RAs will oversee the coordination and monitoring of the overall study. They will prepare all documents required for informed consent and questionnaire administration. They will also be responsible for recruitment, data management (Qualtrics), data analysis, and preparation of presentations and manuscripts. They will be trained on the TTO, VFQ-25, CES-D, HADS-A, PSQI, and CIQ by the Primary Investigator (PI). They will receive ongoing supervision throughout the study by the PI and the co-investigator with the aim of approaching a reliability level of Intra Class Correlation (ICC) > .80 on all scales. Weekly meetings will be organized by the investigators to ensure recruitment and progression of the study.

Fidelity of Assessments

The RAs will be trained and supervised weekly by the PI.

Recruitment, Screening, and Consent Process

425 eye disease patients will be recruited for this study as described previously in the recruitment procedures section. Physicians at Ivey Eye Institute will identify potential participants based on the inclusion and exclusion criteria, as described previously. The potential participants will be asked whether they wish to participate in the following study. Physicians will then refer the patients expressing interest who meet recruitment criteria to the research assistant (RA) for an in-person interview to obtain informed consent or obtain contact information to obtain informed consent electronically.

Potential participants will be presented with an electronic letter of information and consent (LOI). The RA will briefly describe the study to these potential participants and offer to send an electronic copy of the LOI by e-mail. The LOI will contain the contact information of the study investigators and RAs on the front cover page and the study description. In addition, those patients expressing interest will be asked if they consent to providing their contact information (name, phone number, and/or e-mail address). Upon receiving consent to participate in the study, the RA will collect the participant's email and telephone number and present the online survey to be completed.

If the participant presents significant distress (severe depression as confirmed by a CES-D ≥ 24), the PI will be required to respond within 48 hours upon receiving the questionnaire result. The participant in distress will be referred to a mental health provider for further screening for presence of imminent suicidality and safety. The mental health provider will determine whether they have suicidal intent (the wish to harm or kill themselves). In the rare event that there is what is considered an imminent risk, such participants will be referred to the Centralized Emergency Psychiatry Service (CEPS) at the Victoria Hospital.

OUTCOMES

Main Outcomes

Primary Outcomes

Building an evidence base to provide decision-makers with high quality, timely, and relevant evidence, and translating this knowledge into clinical practices.

Study success criteria: If investigators are able to a) screen at least ten patients per week, (b) at least 60% of eligible patients will be recruited, (c) there will be no more than 30% attrition rate, and additionally if (d) 95% of recruited subjects complete 100% study questionnaires; then study would have been successful.

Secondary Outcomes

Health-Related Quality of Life

Improvement in Health-Related Quality of Life (HRQOL) score as measured by the Time Trade-Off questionnaire (TTO).

Vision-Related Quality of Life

Vision-Related Quality of Life (VRQOL) score as measured by the Visual Function Questionnaire (VFQ-25).

Depression

Depressive symptoms as measured by in Center for Epidemiologic Studies - Depression (CES-D) scores (< 16).

Anxiety

Anxiety symptoms as measured by the Hospital Anxiety and Depression Scale - Anxiety subscale (HADS-A) scores

Sleep Quality

Sleep quality as measured by reduction in Pittsburgh Sleep Quality Index (PSQI) scores (≤ 5).

Community Integration

Enhanced community integration as measured by an increase in Community Integration Questionnaire (CIQ) scores.

Qualitative Measures Outcomes

Mental health, physical health, patient experience with virtual care, fear of vision loss, and change in vision during the pandemic as measured using 5-point Likert scale multiple-choice format questionnaires.

STATISTICAL ANALYSIS AND SAMPLE SIZE

Data analysis

The investigators will examine the descriptive statistics for the participants group and check for outliers. It is planned to use a linear-mixed model with the score as the dependent variable, demographic variables as covariates. Univariate and bivariate analysis will be performed for each independent variable against the dependent variable to elicit the impact of each co-variate on the pattern of preference based HRQoL, depression, anxiety, community integration, and sleep quality without adjusting for the effect of other variables. Models will be deemed statistically significant if they are associated with a significant F value (p < 0.01) and if they explain over 15% variability of the dependent variable. Only those independent variables that are statistically significantly associated with the preference based HRQoL (p < 0.05) will be used for model construction.

STATA 15.0 will be used to run all statistical analysis. Based on population size of adults with eye diseases above the age of 65 in South Western Ontario, 5% margin of error, and 95% confidence interval, the sample size has been computed to be 384 participants. Given a 10% attrition rate, the study sample size of 425 participants will be adequate. As such, the sample size has been set to n = 425.

POTENTIAL RISKS/ADVERSE EFFECTS

Risks and Safety of Participants

There are also no direct risks associated with administering the questionnaires to the participants in this study. It does not involve any procedures or medical tests. It is not anticipated that there will be any increased risk in completing any of the questionnaires. It could be that certain questionnaire items make one remember life events which could be potentially disconcerting. Any indications of serious mental health issues will be reported immediately for further clinical assessment and management. Standard of care will be unaffected and only capable and consenting participants will be recruited into the study. COVID-19 restrictions will be respected including the proper donning of personal protective equipment, and sanitation of surfaces and hands. Potential risks to data collection include a privacy breach since there will be various questionnaires to collect information from patients.

Privacy, Confidentiality, and Data Protection

Electronic research records will be stored using QUALTRICS up to a period of 15 years. Study team members may access data on QUALTRICS, download this data and store the data. Any such activities will be done under the direction and supervision of the PI. Data will be coded to protect participant confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with an eye disease by an experienced ophthalmologist.
* Patients with eye diseases age 65 and above.
* Be able to provide valid informed consent to participate in the research study.
* Being able to read and understand English.
* Having no significant self-reported or a physician diagnosed mental health disorder.

Exclusion Criteria:

* Inability to provide a valid informed consent.
* Significant communication barriers or lack of English proficiency that prevents participants from completing the questionnaires.
* Severe depression as confirmed by a CES-D ≥ 24.
* Having a lifetime diagnosis of self-reported other serious mental disorders, including bipolar I or II disorder, primary psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder).
* Self-reported substance abuse or dependence within the past 3 months.
* Having an acutely unstable medical illnesses, including delirium or acute cerebrovascular or cardiovascular events within the last 6 months.
* Having irreversible vision loss that prevents one from completing the questionnaires.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients from the Ivey Eye Institute, St. Joseph's Health Care London, ON will be recruited in-person based on inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
health-related quality of life (HRQoL) | Immediately upon receiving the participant's consent to participate in the study
  HRQoL is an essential measure of quality of life related to health; it helps physician identify hidden morbidity in clinical care as well as improves patient-physician communications. HRQoL will be measured using time trade-off questionnaire. It is measured in a scale of 0 to 1, with higher scores indicating a better outcome. This means that 0 indicates poor HRQoL and 1 indicates perfect health.

SECONDARY OUTCOMES:
Visual Function Score | Immediately upon receiving the participant's consent to participate in the study
  Visual Function score will be measured using Visual Function Questionnaire (VFQ-25). It is measured in a scale of 0 to 100, with 100 indicating the best possible outcome. This means that 0 indicates poor vision-related QOL and 1 indicates perfect health.
Depression | Immediately upon receiving the participant's consent to participate in the study
  Depression is a feeling of severe despondency and dejection. Depression will be measured using the Center for Epidemiological Studies - Depression (CES-D) score. It is measured in a scale of 0 to 60, with higher scores indicating a worse outcome. This means that 0 indicates perfect health and 60 indicates severe depression.
Anxiety | Immediately upon receiving the participant's consent to participate in the study
  Anxiety will be measured using Hospital Anxiety and Depression Scale - Anxiety (HADS-A) subscale. It is scored on a scale of 0 to 21, with higher scores indicating a worse outcome. This means that 0 indicates perfect health and 21 indicates severe anxiety.
Sleep Quality | Immediately upon receiving the participant's consent to participate in the study
  Sleep quality as measured using the Pittsburgh Sleep Quality Index (PSQI) scores. It is scored in a scale of 0 to 21, with higher scores indicating a worse outcome. This means that 0 indicates perfect health and 21 indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Monali Malvankar, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The code key with identifying data (ID #, phone #, date of birth, date of first assessment/consent, date of exit from the study, and any adverse events) will be stored in a password-protected and encrypted spreadsheet on the hospital network shared drive.
  We do not anticipate the questionnaire data collection to take longer than 12 months, and do not anticipate data analysis to take longer than 12 months thereafter (total of 12 months' time), with an absolute maximum of 15 years in post study completion prior to destruction of the data.

REFERENCES:
- [Background] Globe DR, Varma R, Torres M, Wu J, Klein R, Azen SP; Los Angeles Latino Eye Study Group. Self-reported comorbidities and visual function in a population-based study: the Los Angeles Latino Eye Study. Arch Ophthalmol. 2005 Jun;123(6):815-21. doi: 10.1001/archopht.123.6.815. PMID 15955983
- [Background] Sabel BA, Wang J, Cardenas-Morales L, Faiq M, Heim C. Mental stress as consequence and cause of vision loss: the dawn of psychosomatic ophthalmology for preventive and personalized medicine. EPMA J. 2018 May 9;9(2):133-160. doi: 10.1007/s13167-018-0136-8. eCollection 2018 Jun. PMID 29896314
- [Background] Salari N, Hosseinian-Far A, Jalali R, Vaisi-Raygani A, Rasoulpoor S, Mohammadi M, Rasoulpoor S, Khaledi-Paveh B. Prevalence of stress, anxiety, depression among the general population during the COVID-19 pandemic: a systematic review and meta-analysis. Global Health. 2020 Jul 6;16(1):57. doi: 10.1186/s12992-020-00589-w. PMID 32631403
- [Background] Lam DSC, Wong RLM, Lai KHW, Ko CN, Leung HY, Lee VYW, Lau JYN, Huang SS. COVID-19: Special Precautions in Ophthalmic Practice and FAQs on Personal Protection and Mask Selection. Asia Pac J Ophthalmol (Phila). 2020 Mar-Apr;9(2):67-77. doi: 10.1097/APO.0000000000000280. PMID 32349113
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Aylward, Bruce (WHO); Liang, W. (PRC). Report of the WHO-China Joint Mission on Coronavirus Disease 2019 (COVID-19). 2020; vol. 2019 16-24.
- [Background] Quillen DA. Common causes of vision loss in elderly patients. Am Fam Physician. 1999 Jul;60(1):99-108. PMID 10414631